CLINICAL TRIAL: NCT04316104
Title: CuidaTXT: a Text Message Dementia-caregiver Intervention for Latinos
Acronym: CuidaTXT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00144478; 1R21AG065755-01A1 (NIH)
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Caregiver Burnout
Keywords: Dementia; Caregiver; mHealth; Stress; Latino; Disparities
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Intervention Model Description: This intervention, CuidaTXT [Spanish for self-care and texting], will be available in English and Spanish, incorporate two-way messaging and will tailor text messages to the preferences of Latino caregivers. CuidaTXT will be multicomponent and based on the Stress Process Framework as supported by evidence. The intervention will incorporate social support and coping components including dementia education, problem-solving skills training, social network support, care management and referral to community resources.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CuidaTXT (Experimental): This intervention, CuidaTXT [Spanish for self-care and texting], will be available in English and Spanish, incorporate two-way messaging and will tailor text messages to the preferences of Latino caregivers. CuidaTXT will be multicomponent and based on the Stress Process Framework as supported by evidence. The intervention will incorporate social support and coping components including dementia education, problem-solving skills training, social network support, care management and referral to community resources.
  Interventions: Behavioral: CuidaTXT

INTERVENTIONS:
Behavioral: CuidaTXT — Culturally tailored text messages including dementia education, problem-solving skills training, social network support, care management and referral to community resources.

SUMMARY:
Latino families with dementia experience substantial disparities in access to caregiver support compared to their non-Latino white peers, putting them at an increased risk for negative emotional, physical and financial outcomes. This R21 will address this research gap by 1) Developing a culturally and linguistically appropriate text message intervention for caregiver support among Latino family caregivers of individuals with dementia and 2) Testing the feasibility and acceptability of CuidaTXT, a multicomponent text message caregiver support intervention culturally and linguistically tailored for the Latino community.

DETAILED DESCRIPTION:
Latino relatives of individuals with dementia are less likely than non-Latino whites to have access to caregiver support. Text messaging can dramatically enhance the reach of effective culturally and linguistically tailored caregiver support interventions. However, to our knowledge, no text message interventions exist to provide caregiver support among caregivers of individuals with dementia. Text message interventions can capitalize on the fact that Latinos own cellphones and use them to text at a higher rate than non-Latino whites. The overall aim of this proposal is to develop and test the first text message intervention for caregiver support of individuals with dementia among Latinos. This intervention, CuidaTXT [Spanish for self-care and texting], will be available in English and Spanish, incorporate two-way messaging and will tailor text messages to the preferences of Latino caregivers. CuidaTXT will be multicomponent and based on the Stress Process Framework as supported by evidence. The intervention will incorporate social support and coping components including dementia education, problem-solving skills training, social network support, care management and referral to community resources. This research corresponds with Stage 1 of the NIH Stage Model for Behavioral Intervention Development. In Aim 1, researchers will develop a culturally and linguistically appropriate text message intervention for caregiver support among Latino family caregivers of individuals with dementia using user-centered design methods. In Aim 2, researchers will test the feasibility and acceptability of CuidaTXT during six months.

ELIGIBILITY:
Inclusion Criteria:

* Spanish and English-speaking individuals
* Over the age of 18
* Identify as Latino
* Report providing hands-on care for a relative who has been given a clinical or research dementia diagnosis
* Care recipient has an AD-8 screening score greater than or equal to 2, indicating cognitive impairment
* Self-report being able to read and write
* Self-report owning a cell phone with a flat fee and use it at least weekly for texting

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include caregivers' demographic and behavioral data from interviews as well as metrics, direct observation and survey data on feasibility, acceptability and preliminary efficacy of CuidaTXT. Along with the dataset, the team will create a code book documenting all variables. Although the data analytic files will not have direct identifiers (only study identification numbers), the possibility of deductive disclosure of subjects with certain clinical characteristics may remain. To safeguard against the unlikely event of deductive disclosure, the team will only make the data files and codebook available to other researchers on a case-by-case basis.
Supporting Information: Analytic Code
Time Frame: Data will become available on July 1st, 2022
Access Criteria: Researchers requesting data will need to complete a request form outlining intended use of the data, and agree to use the data solely for this intended purpose. Prior to data release, researchers requesting data will be required to sign a confidentiality agreement specifying that they will not identify any individual participant, that they will use secure technology to safeguard the data, and that they will destroy or return the data after their analyses are completed.

RESULTS

PARTICIPANT FLOW:
Groups:
- CuidaTXT: This intervention, CuidaTXT [Spanish for self-care and texting], will be available in English and Spanish, incorporate two-way messaging and will tailor text messages to the preferences of Latino caregivers. CuidaTXT will be multicomponent and based on the Stress Process Framework as supported by evidence. The intervention will incorporate social support and coping components including dementia education, problem-solving skills training, social network support, care management and referral to community resources.
  CuidTXT: Culturally tailored text messages including dementia education, problem-solving skills training, social network support, care management and referral to community resources.
Period: Overall Study
Arm/Group | CuidaTXT
Started | 24
Completed | 21
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- CuidTXT: This intervention, CuidaTXT [Spanish for self-care and texting], will be available in English and Spanish, incorporate two-way messaging and will tailor text messages to the preferences of Latino caregivers. CuidaTXT will be multicomponent and based on the Stress Process Framework as supported by evidence. The intervention will incorporate social support and coping components including dementia education, problem-solving skills training, social network support, care management and referral to community resources.
  CuidTXT: Culturally tailored text messages including dementia education, problem-solving skills training, social network support, care management and referral to community resources.
Arm/Group | CuidTXT
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 2
  Unknown or Not Reported | 15
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Able to Opt Into CuidaTXT (Enrollment Feasibility)
Description: Metrics of the percentage of participants able to opt into CuidaTXT. Each participant the researcher is able to enroll into the CuidaTXT intervention via entering their name and phone number in the software is counted here. The result of being enrolled successfully is that the participant reports receiving text messages to the research team during the call when the enrollment takes place. Participants for whom the name and phone number is not able to be entered in the software, or who report not receiving text messages upon entering their information in the software are not counted, as this would be an unsuccessful attempt of enrollment into CuidaTXT.
Time Frame: During the 6 months of the intervention period
Measure: Count of Participants; unit: Participants
Arm/Group | CuidTXT
Number analyzed (Participants) | 24
Participants | 24

2. Primary Outcome: Percentage of Participants Who Texted the STOP Keyword to Opt Out/Quit the Intervention
Description: Metrics of percentage of participants who texted STOP keyword. Participants are instructed during the course of the intervention to send the keyword STOP if they want to quit the intervention. The research team counts each participant who sends the keyword STOP, as seen on the software report, and calculates a percentage among all the participants.
Time Frame: During the 6 months of the intervention period
Measure: Count of Participants; unit: Participants
Arm/Group | CuidTXT
Number analyzed (Participants) | 24
Participants | 0

3. Primary Outcome: Number of Participants Who Reported Experiencing Technical Problems With the Intervention
Description: Survey open-ended reports of technical problems. A question in the 6 month survey asks whether participants experienced any technical problems with CuidaTXT during the study. The response options are Yes or No. The outcome is the number of participants who responded Yes to this question among all the participants who completed the 6 month survey.
Time Frame: 6 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | CuidTXT
Number analyzed (Participants) | 21
Participants | 2

4. Primary Outcome: Percentage of Participants Who Interacted With the Intervention by Sending at Least One Text Message (Engagement Feasibility)
Description: Metrics on percentage of participants who sent at least one text message. The CuiaTXT intervention consists of participants receiving and sending messages to the program. The research team has access to the CuidaTXT software, where they can see the messages each participant has sent to the program. This metric is the number of participants who sent at least one text message to CuidaTXT among all the participants.
Time Frame: During the 6 months of the intervention period
Measure: Count of Participants; unit: Participants
Arm/Group | CuidTXT
Number analyzed (Participants) | 24
Participants | 22

5. Primary Outcome: Thoroughness With Which Participants Read Intervention Text Messages (Engagement Feasibility)
Description: Survey responses of percentage of participants who report reading most or all texts thoroughly. The 6 month survey asks participants to what extent they have read the text messages. There are 3 response options: 'I read through the text messages thoroughly most times' in the follow-up survey as opposed to 'I took only a short look at the text messages most times', or 'I did not read the text messages most times'. The current outcome indicates the number of participants who responded 'I read through the text messages thoroughly most times' among all participants that completed the 6 month survey.
Time Frame: 6 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | CuidTXT
Number analyzed (Participants) | 21
Participants | 18

6. Primary Outcome: Average of the Percentage of Messages Sent by Each Participant to Interact With the Intervention That Were Keywords
Description: Metrics of the percentage of messages sent by participants to interact with the intervention that were keywords. Participants were able to send text messages to receive tailored text messages back about topics to cover their needs. Text messages they could send include chat messages with a live coach (e.g., like any text message people send ordinarily) or keyword-driven messages (a specific keyword that triggers an automatic message). The research team counted the number of messages in the software report that were keywords and chat messages and calculated the percentage of those that were keywords and later calculated the average of that percentage for all participants.
Time Frame: During the 6 months of the intervention period
Measure: Mean (Standard Deviation); unit: Percent of messages were keywords
Arm/Group | CuidTXT
Number analyzed (Participants) | 24
Percent of messages were keywords | 44.1 (30.6)

7. Primary Outcome: Satisfaction With Intervention
Description: Research team-developed one item with a 4-item Likert scale on satisfaction with intervention, higher scores meaning higher satisfaction. In the 6 month survey, participants were asked what their levels of satisfaction are regarding the intervention as a whole. Options ranged from Not at All (1) to Extremely (4).
Time Frame: 6 months from baseline
Population: Average satisfaction score in a 1-item scale that ranges from Not at All (1) to Extremely (4) satisfied.
Measure: Mean (Standard Deviation); unit: Average score
Arm/Group | CuidTXT
Number analyzed (Participants) | 21
Average score | 3.6 (0.5)

8. Secondary Outcome: Change From Baseline to 6 Months in Alzheimer's Disease Knowledge
Description: Epidemiology/Etiology Disease Scale: 14-item, true/false scale takes approximately 5-10 min to complete. An example of an item is "There is no cure for Alzheimer's". Each correct answer is scored as 1 point and each incorrect answer as 0 points. Points are summed up for a total score, which ranges from 0 to 14. Higher scores mean more questions answered correctly. The current outcome is the scales' score at month 6 minus the score at baseline.
Time Frame: Baseline and 6 months from baseline
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | CuidTXT
Number analyzed (Participants) | 21
change in units on a scale | 1.1 (1.7)

9. Secondary Outcome: Change From Baseline to 6 Months in Caregiver Social Support
Description: Interpersonal Support Evaluation List-12 (ISEL-12): 12-item instrument that that yields a total score that describes overall perceived social support, and three subscales representing perceived availability of appraisal (advice or guidance), belonging (empathy, acceptance, concern), and tangible (help or assistance, such as material or financial aid) social support. Each item is rated either definitely false (1), probably false (2), probably true (3), or definitely true (4). Scores are summed for the total scale (12-48) and subscales (4-16). Higher scores mean higher social support for each scale. The current outcome is the scales' score at month 6 minus the score at baseline.
Time Frame: Baseline and 6 months from baseline
Measure: Mean (Standard Deviation); unit: Change in units of scale
Arm/Group | CuidTXT
Number analyzed (Participants) | 20
Change in units of scale | 1.0 (3.2)

10. Secondary Outcome: Change From Baseline to 6 Months in Caregiving Self-efficacy
Description: Preparedness for caregiving scale: The Preparedness for Caregiving Scale is a caregiver self-rated instrument that consists of eight items that asks caregivers how well prepared they believe they are for multiple domains of caregiving. Preparedness is defined as perceived readiness for multiple domains of the caregiving role such as providing physical care, providing emotional support, setting up in-home support services, and dealing with the stress of caregiving. Responses are rated on a 5 point scale with scores ranging from 0 (not at all prepared) to 4 (very well prepared). The total score is the sum of all items divided by the number of items (eight), and ranges from 0 to 4. The higher the score the more prepared the caregiver feels for caregiving. An example of an item is: "How well prepared do you think you are to take care of your family member's physical needs?". The current outcome is the scales' score at month 6 minus the score at baseline.
Time Frame: Baseline and 6 months from baseline
Measure: Mean (Standard Deviation); unit: Change in units of scale
Arm/Group | CuidTXT
Number analyzed (Participants) | 20
Change in units of scale | 0.5 (0.5)

11. Secondary Outcome: Change From Baseline to 6 Months in Caregiver Depression
Description: 10-item Center for Epidemiologic Studies-Depression scale (CES-D-10): This is a 10-item, self-report rating scale that measures characteristic symptoms of depression in the past week (e.g. depression, loneliness, restless sleep). Each item is rated on a 4-point scale, from 0 (rarely or none of the time) to 3 (most or all of the time) with positively worded items (items 5 and 8) reverse scored. Items yield summary scores that range from 0 to 30, with higher scores indicating higher severity. An example of an item is: "I was bothered by things that usually don't bother me". The current outcome is the scales' score at month 6 minus the score at baseline.
Time Frame: Baseline and 6 months from baseline
Measure: Mean (Standard Deviation); unit: Change in units of scale
Arm/Group | CuidTXT
Number analyzed (Participants) | 20
Change in units of scale | -3.4 (5.2)

ADVERSE EVENTS:
Time Frame: 6 months
Description: No systemic assessment of adverse events was used
Arm/Group | CuidTXT
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT04316104/Prot_SAP_ICF_000.pdf